CLINICAL TRIAL: NCT01256372
Title: An Explorative Phase 2, Randomized, Double-Blind, Placebo-Controlled, Safety and Efficacy Trial of Two Dosing Regimens of AP214 for the Prevention of Kidney Injury in Patients Undergoing Cardiac Surgery
Brief Title: An Trial of Two Dosing Regimens of AP214 for the Prevention of Kidney Injury in Patients Undergoing Cardiac Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Action Pharma A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AP214-CS007
Record Dates: First submitted 2010-12-05; First posted 2010-12-08 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Cardiac Surgery; Coronary Artery Bypass; Aortic Aneurysm; Valve Surgery; Kidney Diseases
Keywords: Cardiac surgery; Acute kidney injury
MeSH Terms: conditions — Aortic Aneurysm; Kidney Diseases; Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- AP214; dose-level 1 (Experimental): AP214; dose-level 1
  Interventions: Drug: AP214
- AP214; dose-level 2 (Experimental): AP214; dose-level 2
  Interventions: Drug: AP214
- Placebo to AP214 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AP214 — AP214
  Arms: AP214; dose-level 1; AP214; dose-level 2
Drug: Placebo — Placebo; intravenous infusion
  Arms: Placebo to AP214

SUMMARY:
This study investigates the effect of two dose-levels of AP214 on the prevention of (acute) kidney injury after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Has signed the trial-specific informed consent form.
2. Patients ≥ 18 years old, male or female, not of childbearing potential (postmenopausal or permanently sterilized, e.g. tubal ligation, hysterectomy, bilateral salpingectomy), regardless of ethnicity.
3. Patients undergoing combined coronary artery bypass grafting (CABG) surgery and surgery of one or more cardiac valve (valve(s) surgery), or
4. Patients undergoing surgery of more than one cardiac valve (valves surgery), or
5. Patients undergoing surgery of the aortic root or ascending part of the aorta, or
6. Patients undergoing surgery of the aortic root or ascending part of the aorta, combined with CABG and/or valve(s) surgery, or
7. Patients with stage III chronic kidney disease (eGFR 30-59 ml/min determined by the Modification of Diet in Renal Disease (MDRD formula)) undergoing CABG or Valve surgery

Exclusion Criteria:

1. Cardiac surgery to be performed "off pump" without cardiopulmonary bypass.
2. Cardiac surgery to be performed with hypothermic circulatory arrest.
3. Confirmed or suspected endocarditis.
4. EF ≤ 20%, evaluated within 2 months prior to screening visit.
5. Requiring a reoperation on one of the valves within 3 months following the original valve surgical procedure.
6. Active peptic ulcer disease and gastritis.
7. Receiving dopamine, adrenalin or noradrenalin at any dose at any time 14 days prior to Day of surgery.
8. Known or suspected hypersensitivity to the investigational medicinal product.
9. Current participation in any other interventional clinical trial.
10. Previously dosed with AP214.
11. Use of investigational medicinal products within the previous 6 months.
12. Body weight above 130 kg.
13. History of any organ transplant.
14. Women who are of childbearing potential, pregnant, or breast-feeding.
15. Current abuse of alcohol or substance, according to the investigator's medical judgment.
16. Has a mental incapacity or language barriers precluding adequate understanding of trial procedures.
17. Any history of cancer within the last 2 years
18. Any history of dialysis.
19. Is considered by the Investigator unsuitable to participate in the trial for any other reason, for instance due to a significant serious underlying condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | 90 days
  To assess the safety and tolerability of AP214 compared to placebo; by analysis of number and nature of Adverse Events (AEs), Serious Adverse Events (SAEs), changes in laboratory parameters and overall health status
Efficacy | 7 days
  To assess the effect of AP214 versus placebo on the maximal postoperative change in absolute values of Serum Creatinine (SCr) compared to baseline within the first 7 days after surgery or until discharge from hospital, whichever comes first

SECONDARY OUTCOMES:
Efficacy | 90 days
  To assess the ability of AP214 compared to placebo to reduce postoperative changes in SCr, and eGFR at day 28, 60 and Day 90 and GFR at Day 90 compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Action Pharma, Study Director — Action Pharma A/S
Locations (1):
- University Hospital Copenhagen, Rigshospitalet, Copenhagen, Denmark